CLINICAL TRIAL: NCT07148245
Title: Characterization of the Symptom Experience of Patients With Cutaneous Melanoma Receiving Immune Checkpoint Inhibitor Therapy
Brief Title: Symptoms of Immune Checkpoint Inhibitor Therapy in Cutaneous Melanoma
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 25858; NCI-2025-05718 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); 4R00CA286967 (NIH)
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Cutaneous Melanoma; Cutaneous Melanoma, Stage III; Cutaneous Melanoma by AJCC V7 Stage; Cutaneous Melanoma, Stage IV
Keywords: Toxicity
MeSH Terms: conditions — Melanoma | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be obtained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults treated with Immune Checkpoint Inhibitor Therapy: Adult participants diagnosed with stage IIB to IV cutaneous melanoma who will begin immune checkpoint therapy at University of California, San Francisco medical center locations.
  Interventions: Procedure: Blood Sample; Other: Health Related Quality of Life Questionnaires (HRQoL); Other: Medical Chart Review

INTERVENTIONS:
Procedure: Blood Sample — Blood samples will be collected
Other: Health Related Quality of Life Questionnaires (HRQoL) — Participants may be given HRQoLs during the course of data collection
  Other Names: Quality of Life Questionnaires; Surveys
Other: Medical Chart Review — Participants will undergo medical charts review during the course of data collection
  Other Names: Chart review

SUMMARY:
The introduction of immune checkpoint inhibitors (ICIs) for the treatment of patients with stages IIB to IV cutaneous melanoma resulted in dramatic improvements in mortality rates for this common form of cancer. With this rapid shift in treatment, significant gaps in knowledge exist regarding the impact of ICIs on patients' symptom experiences. An in-depth characterization of inter-individual differences in patients' symptom experiences will fill this knowledge gap and assist with the early detection of ICI toxicity; guide symptom management; inform treatment decision making; and refine ICI-symptom instrument development. Furthermore, given the limited knowledge in this area, the identification of demographic, clinical, environmental, and molecular risk factors associated with a worse symptom experience is warranted. This is a longitudinal, prospective study evaluating the symptoms that immune checkpoint inhibitors may cause in patients with cutaneous melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. Evaluate for changes over time in the patients' symptom experience,
2. Identify distinct symptom profiles over time.
3. Evaluate for demographic, clinical, environmental, and molecular risk factors associated with a worse profile.

OUTLINE:

Participants receiving ICI outside the scope of this study as part of usual care will have a chart review from the first cycle of non-investigational treatment for up to 4 cycles. Participants may complete symptom and health-related quality of life questionnaires during the course of the study, and blood samples will be obtained at regular clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Able to speak and read English
* Diagnosed with stage IIB, III, or IV cutaneous melanoma
* Participants who are scheduled to receive >=1 immune checkpoint inhibitor at University of California San Francisco medical center locations. Participants on targeted therapies (e.g., BRAF or mitogen-activated extracellular signal-regulated kinase (MEK) inhibitors) will be eligible.
* Provide written informed consent to participate in this study.
* Participants with stage IIB or higher cutaneous melanoma

Exclusion Criteria:

* Participants will be excluded if they are unable to complete study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with stage IIB, III, or IV cutaneous melanoma who will receive ≥ 1 immune checkpoint inhibitor therapy as part of treatment for cutaneous melanoma.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of symptoms reported over time | Up to 5 months
  Evaluations of symptoms over time will be assessed via calculating the occurrence rates and means and standard deviations for the severity and distress ratings for all 53 symptoms and determine the most common, severe, and distressing symptoms over time.
Number of distinct symptom profiles identified | Up to 5 months
  Latent class analysis will be used to identify subgroups of patients with distinct symptom occurrence profiles separately at each time point. Only symptoms that occurred in ≥20% of patients will used in the latent class analysis.
Number of risk factors identified with worse symptom profile over time. | Up to 5 months
  Associations among the latent symptom occurrence profiles in demographic, clinical, environmental, and molecular characteristics along with financial toxicity, quality of life, and cancer-related distress will be evaluated using parametric and non-parametric methods to identify risk factors associated with a worse symptom profile over time.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Harris, PhD, RN, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets may be shared with study collaborators during the course of the study.
Supporting Information: Study Protocol, SAP, ICF